CLINICAL TRIAL: NCT07170137
Title: Comparison of Uterine Distension in Hysterosonography Among Patients Monitored for Infertility
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0112.1_PMA
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Infertile Women Undergoing IVF or ICSI; Distension by Volumetric Analysis of the Uterus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- infertile women
- fertile women

SUMMARY:
Comparison of differences in distension by volumetric analysis of the uterus before and after distension between groups of infertile and apparently fertile women.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 18 and < 43 years old
* No contraindications to pregnancy
* Patients consulting at the Saint Denis assisted reproductive technology (ART) department due to desire to become pregnant or infertility

Exclusion Criteria:

* Contraindication to assisted reproductive technology treatment

Ages: 18 Years to 43 Years | Sex: Female
Age Groups: Adult
Study Population: women seeking assisted reproductive technology (ART)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
uterine distension | 1 years

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier Delafontaine, Saint-Denis, France